CLINICAL TRIAL: NCT06939998
Title: A Nontraditional Approach for Awake Fiberoptic Nasotracheal Intubation. A Randomized Controlled Superiority Trial
Brief Title: A Nontraditional Approach for Awake Fiberoptic Nasotracheal Intubation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRP number 00012098
Record Dates: First submitted 2025-03-04; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-01

CONDITIONS: Endotracheal Tube Placement
Keywords: nasotracheal fiberoptic intubation through ETT

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CFOBI conventional fiberoptic intubation (Experimental): a 5.0-mm flexible fiberoptic bronchoscope (Pentax) will be loaded with an endotracheal tube of the proper size (7.5 for male and 7.0 for female patients). The bronchoscope tip will then be introduced into the nasal cavity, and the vocal cords will be detected.
  Interventions: Procedure: CFOBI
- FOBIET nasotracheal fiberoptic intubation through an endotracheal tube in the nasopharynx (Active Comparator): FOBIET: an endotracheal tube (ET) is initially inserted into the nasal cavity, and then a flexible fiberoptic bronchoscope is introduced through it. The endotracheal tube will be connected to a catheter mount by which the investigator can deliver oxygenation. When using a nasal endotracheal tube, the tip is lubricated with 2% lignocaine jelly before being inserted into the nasal cavity and pushed up and down to allow the jelly to spread. The fiberoptic bronchoscope descends through the endotracheal tube after being inserted into the nasal passage as a nasal airway in the direction of the vocal cords until they can be seen
  Interventions: Procedure: FOBIET

INTERVENTIONS:
Procedure: FOBIET — an endotracheal tube (ET) is initially inserted into the nasal cavity, and then a flexible fiberoptic bronchoscope is introduced through it. The endotracheal tube will be connected to a catheter mount by which the investigator can deliver oxygenation. When using a nasal endotracheal tube, the tip is lubricated with 2% lignocaine jelly before being inserted into the nasal cavity and pushed up and down to allow the jelly to spread. The fiberoptic bronchoscope descends through the endotracheal tube after being inserted into the nasal passage as a nasal airway in the direction of the vocal cords until they can be seen.
  After identifying the vocal cords, 2 ml of 2% lidocaine will be sprayed over the supraglottic area using the bronchoscope's working channel. An additional 2 ml of 2% lidocaine will then be sprayed directly onto the vocal cords, after which the tip of an endotracheal (ET) tube will be carefully inserted into them.
  Other Names: fiberoptic intubation through nasal endotracheal tube
  Arms: FOBIET nasotracheal fiberoptic intubation through an endotracheal tube in the nasopharynx
Procedure: CFOBI — a 5.0-mm flexible fiberoptic bronchoscope (Pentax) will be loaded with an endotracheal tube of the proper size (7.5 for male and 7.0 for female patients). The bronchoscope tip will then be introduced into the nasal cavity, and the vocal cords will be detected.
  Arms: CFOBI conventional fiberoptic intubation

SUMMARY:
The goal of this clinical trial is to learn if awake nasotracheal fiberoptic intubation through an endotracheal tube inserted in the nasopharynx would be quick and have fewer complications than the conventional technique. The main questions it aims to answer are:

which technique of intubation is faster, with more patient comfort and satisfaction? which technique has fewer complications like cough, bleeding, and laryngospasm? Researchers will compare intubation with the conventional fiberoptic technique for intubation to awake nasotracheal fiberoptic intubation through an endotracheal tube inserted in the nasopharynx.

Participants will be monitored throughout the procedure for:

1. The duration of the intubation procedure
2. The mean peripheral oxygen saturation
3. Hemodynamic variables (HR, MAP)

DETAILED DESCRIPTION:
A nontraditional approach for awake fiberoptic nasotracheal intubation. A randomized controlled superiority trial Introduction It takes skill and specialized equipment to intubate someone with an anticipated difficult airway. The American Society of Anaesthesiologists and other European authors advise awake fiberoptic intubation (FOB). An awake patient can protect the airway. When a patient breathes independently until the airway is secured, awake fiberoptic intubation increases safety. In addition to requiring awake flexible fiberoptic intubation, difficult airway instances such as limited jaw mobility, restricted mouth opening, surgical interventions, or procedures planned in the oral cavity also require the nasotracheal route for intubation. Compared to oral intubation, nasal intubation is typically more straightforward and more successful.

Negotiating the endotracheal tube can be challenging since initial resistance is experienced during the passage of the bronchoscope and endotracheal tube (ET). However, the nasal approach gives an aligned airway to the larynx and trachea and holds the tube more stably. Gentle force is needed to overcome this resistance, which could cause the nose passage's friable mucosa to bleed. Coughing during a flexible fiberoptic bronchoscopy can make it difficult to see the vocal cord because bleeding in the nasopharynx and oropharynx can irritate the airway and cause coughing.

Berman and Ovassapian airways are available to help with awake flexible fiberoptic intubation via oral route. These airways provide a passageway for the ET tube and bronchoscope. However, the nasal approach does not have access to such an airway. A fiberoptic bronchoscope is usually passed through the more patent nostril to reach the nasopharynx. It then follows the main nasal pathway at the nose floor along the superior aspect of the hard palate and the lateral aspect of the nasal septum inferior to the lower turbinate. Once there, the operator can identify the pharyngeal structures, such as the base of the tongue and the epiglottis, which are primarily "in-fall" and prevent clear views of the larynx, necessitating a jaw thrust to visualize the laryngeal structures for patients who are scheduled to be intubated under general anesthesia so a wake fiberoptic is preferred in anticipating difficult airway.

An endotracheal tube (ET) can be inserted along the FOB cable that has already advanced into the trachea, making FOB nasal intubation easier and faster. This is achieved by inserting a modified split tube nasally down to or near the larynx, which allows the FOB cable to be immediately in front of the larynx without the need to confirm the anatomical details of the nasopharyngeal-laryngeal journey required during classic nasal FOB intubation.

This study hypothesized that awake nasotracheal fiberoptic intubation through an endotracheal tube inserted in the nasopharynx would be quick and have fewer complications than the conventional technique. This study compares the time to intubation and safety of FOB nasal intubation as classically done and thorough endotracheal tube.

Objectives The study's primary objective will be to determine the time taken for intubation. Its secondary objectives will be to observe desaturation episodes during the procedure, complications like cough, bleeding, and laryngospasm, and patient comfort and satisfaction.

A single-blind, randomized control superiority trial will be conducted after approval from the institutional ethical committee, and the trial will be registered with the clinical trial registry. The trial will be conducted at Alexandra University Hospital. The selection of patients will be based on inclusion criteria. The study will comply with the principles outlined in the Declaration of Helsinki. After explaining the nature and purpose of the trial, informed consent will be obtained from all participants. Before enrolling the patients, the procedure will be described, and informed consent will be taken for nasotracheal fiberoptic intubation, emergency surgical tracheostomy, delayed extubation, anesthesia, and surgery will be taken from patients.

After assessing the inclusion criteria, 112 patients will be randomized using a computer-generated randomization sequence. These selected patients will be divided into two groups. Group allocation (1:1 allocation ratio) will be done using a sealed envelope technique, and patients will be allocated equally to either group CFOBI (conventional fiberoptic intubation) or group FOBIET (fiberoptic intubation through an endotracheal tube). In the traditional fiberoptic intubation group (N = 56), a flexible fiberoptic bronchoscope is first introduced through the nasal passage. In the study group, an endotracheal tube is introduced in the nasal cavity first, and then a flexible fiberoptic bronchoscope will be introduced.

Interventions:

All patients will be premeditated with midazolam 0.03 mg/kg just before the surgery. Five ml of 2% lignocaine + 1 ml adrenaline will be nebulized over twenty minutes to provide a topical anesthetic. One drop of xylometazoline 0.1% will be administered to each patient's nostrils. Before the treatment, a 10% lignocaine spray would be applied bilaterally in the facial pillars. Both groups' tongue depressors will measure how well the topical anesthetic works. A dose of 0.03 to 0.05 mg/kg of injectable midazolam would be administered, and sedation (with a targeted Ramsay sedation score of 3) will be initiated with an intravenous (IV) injection of 1 microgram per kilogram of loading dexmedetomidine over 10 minutes. More patent nostrils will be selected for the treatment, and nasal patency will be performed.

-In the CFOBI group: a 5.0-mm flexible fiberoptic bronchoscope (Pentax) will be loaded with an endotracheal tube of the proper size (7.5 for male and 7.0 for female patients). The bronchoscope tip will then be introduced into the nasal cavity, and the vocal cords will be detected.

-In the FOBIET group: an endotracheal tube (ET) is initially inserted into the nasal cavity, and then a flexible fiberoptic bronchoscope is introduced through it. The endotracheal tube will be connected to a catheter mount by which the investigators can deliver oxygenation. When using a nasal endotracheal tube, the tip is lubricated with 2% lignocaine jelly before being inserted into the nasal cavity and pushed up and down to allow the jelly to spread. The fiberoptic bronchoscope descends through the endotracheal tube after being inserted into the nasal passage as a nasal airway in the direction of the vocal cords until they can be seen.

After identifying the vocal cords, 2 ml of 2% lidocaine will be sprayed over the supraglottic area using the bronchoscope's working channel. An additional 2 ml of 2% lidocaine will then be sprayed directly onto the vocal cords, after which the tip of an endotracheal (ET) tube will be carefully inserted into them.

Bilateral equal air entry and capnography will verify that the ET tube is correctly positioned in the trachea in both groups after the tube has been successfully passed through the vocal cords and the carina has been identified. The tube will then be secured, and the cuff will inflate.

Measurements:

1. The duration of the intubation procedure will be recorded in minutes, starting from the point at which the scope is inserted into the nares and ending with the ET cuff being inflated.
2. The mean peripheral oxygen saturation (Spo2) will be recorded throughout the process.
3. Hemodynamic variables (HR, MAP) will be recorded at three different time intervals (baseline, at the beginning of the procedure during insertion of the endotracheal tube through the nostril in one group, during fiberscope insertion in the other group, and at the end of the study after confirmation of the endotracheal tube in place).
4. Intubation condition scores will be assessed by vocal cord movement (1 = open, 2 = moving, 3 = closing, 4 = closed), coughing (1 = none, 2 = one gag or cough only, 3 = >1 gag or cough, but acceptable conditions, 4 = unacceptable conditions).
5. intubation comfort score (1=noreaction,2=griming,3=verberal objection,4=defensive movement of hands and head).
6. The airway obstruction score of Downes and Raphaelly. Upper airway respiratory distress is graded as: Absent= (0), Mild=(1-3),Moderate=(4-6),Severe=(≥7).
7. Laryngospasm and bleeding incidence will be noted.

Data Collection:

Data will be collected by trained research personnel, entered into a secure database, and maintained following Good Clinical Practice (GCP) guidelines.

Data Analysis: Statistical analysis will be performed using appropriate tests to compare primary and secondary endpoints.

Sample Size:

The sample size was determined for the primary outcome (time for intubation), aiming to demonstrate the new approach's superiority over the conventional approach. A 30 % reduction in time for intubation (min) between groups was considered clinically relevant. Based on another trial , the investigators assumed a time for intubation of 6.15 ± 3.0 min (in patients who underwent conventional awake fiberoptic intubation). Assuming α=0.05 and power=0.90 for a 30 % difference in time for intubation using a two-sided Χ2 test, the calculated sample size will be 112. The sample size required per group will be 56.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 60 years,
* ASA (American Society of Anesthesiologists) grade I to IV, and an
* indication of awake fiberoptic nasal intubation.

Exclusion Criteria:

* Patients who refuse to undergo the procedure and
* patients with any absolute contraindication for nasal intubation like head trauma, suspected base of skull fractures, nasal mass, or deviated nasal septum

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time taken for intubation. | up to 7 month
  The duration of the intubation procedure will be recorded in minutes, starting from the point at which the scope is inserted into the nares and ending with the ET cuff being inflated.

SECONDARY OUTCOMES:
Number of desaturation episodes | up to 7 month
  The mean peripheral oxygen saturation (Spo2) will be recorded throughout the process and SpO2 below 90% will be considered as a desaturation episode.
Occurrence of airway obstruction. | up to 7 month
  The airway obstruction score of Downes and Raphaelly, will be recorded during the intervention. Upper airway respiratory distress is graded as: Absent= (0), Mild=(1-3),Moderate=(4-6),Severe=(≥7).
Patient comfort | up to 7 month
  intubation comfort score will be recorded during the procedure(1=noreaction,2=griming,3=verbal objection,4=defensive movement of hands and head)
Occurrence of other adverse effects | up to 7 month
  any other complication during intervention will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Islam Elbardan, Dr, Principal Investigator — University of Alexandria
Locations (1):
- Alexandria University, Alexandria, Alexandria Governorate, Egypt